CLINICAL TRIAL: NCT05770999
Title: The Effect of Aromatherapy Application on Pain, Stress and Behaviors of the Newborn
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Harun Özbey, Research Assistant, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2021/04-02
Record Dates: First submitted 2022-10-27; First posted 2023-03-16 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Newborn, Infant, Disease
Keywords: Newborn; Aromatherapy; Pain; Stress; Newborn Behaviors
MeSH Terms: conditions — Disease; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Lavender massage (Experimental): A mixture of 20 cc of sweet almond oil and 1 cc of lavender oil will be used. Sweet almond oil has been used to dilute lavender oil. lavender massage lasted about 10 minutes.
  Interventions: Other: Lavender application
- Lavender bath (Experimental): A mixture of 20 cc bath water and 1 cc lavender oil will be used. lavender bath lasted about 10 minutes.
  Interventions: Other: Lavender application
- Control group (No Intervention): The newborns in the control group did not receive any treatment other than their clinical routines (vital signs monitoring, skin care with sunflower oil, eye and mouth care, changing diapers, changing bed linen, feeding and clinical treatments).

INTERVENTIONS:
Other: Lavender application — Lavender application
  Arms: Lavender bath; Lavender massage

SUMMARY:
This study was planned as a randomized controlled double-blind experimental study to examine the effect of aromatherapy on newborn pain, stress and behaviors. The main questions it aims to answer are:

* Lavender oil massage applied to newborns has an effect on pain, stress and behavior of newborns.
* Lavender oil bath applied to newborns has an effect on pain, stress and behavior of newborns.
* There is a difference between lavender oil massage and lavender oil bath applications applied to newborns in reducing the pain and stress level of the newborn and regulating their behavior.

Randomization method will be used in the determination of the study groups (Lavender massage, lavender bath and control group), and the study group to which the newborns will be included will be determined in the computer environment. Gender, gestational age, postnatal age and body weight will be considered as matching criteria for newborns included in lavender massage, lavender bath and control groups. For ALPS-Neo and ABSS evaluations, 10 minutes (20 minutes in total) of newborns will be recorded with a video camera before and after the study.

DETAILED DESCRIPTION:
Newborns have to receive treatment and care for a long time in the neonatal unit. Newborns admitted to neonatal intensive care units (NICUs) have to cope with stressors such as numerous environmental stimuli (bright light, loud noise, frequent touch, etc.) and repetitive painful interventions when they are not developmentally ready. A care environment devoid of parental contact and stimuli, disturbing the newborn, and encountering stress and excessive stimuli negatively affects the delicate physical condition and immature organ systems of the newborn, and physiological and behavioral stress symptoms can be observed. However, in neonatal units; It is known that there may be many undesirable stimuli such as excessive noise, light, and intense activity in the unit, as well as situations where sensory stimuli such as monotonous sounds, inactivity, and silence from some medical equipment are rare. In these cases, sensory deprivation or sensory overload problems may develop as a result of the decrease or increase in the quality and quantity of sensory stimuli . Precautions should be taken to prevent these problems from occurring. Complementary care practices such as aromatherapy can be used to reduce sensory stimulus problems and stress.

Aromatherapy, which is the most widely used in complementary care applications; It is defined as the use of essential oils obtained from flowers, plants and trees to increase health and well-being. Essential oils can be administered orally, by touch, and by inhalation. The aim of aromatherapy by touch (massage, bath, compress) is to benefit from the anti-inflammatory, antispasmadic, antiviral, antifungal and antibacterial effects of essential oils and to allow the muscles to return to a resting tone. Since the sense of touch is developed in newborn babies at birth, the application of aromatic oils with the sense of touch is important in reducing the stress of the baby in the first days of his life.

Among the essential oils used in aromatherapy, the most studied fragrance is lavender. Lavender generally has antiseptic, anti-inflammatory, pain-relieving, relaxing and sleep-inhibiting effects. In line with this information, it is aimed to examine the effect of aromatherapy on the pain, stress and behavior of newborns.

ELIGIBILITY:
Inclusion Criteria:

* Postnatal age of 1-5 days,
* Gestational age is 38-42 weeks,
* Tolerant of enterally given food (without NEC, digestive system and chromosomal abnormalities),
* Not connected to respiratory support device,
* No skin disease,
* No surgical intervention,
* Newborns with written consent from at least one of the parents will be included in the study.

Exclusion Criteria:

* Findings such as tachypnea, fever
* Newborns with Rh and AB0 incompatibility
* Newborns undergoing surgical intervention

Ages: 1 Day to 5 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2022-05-21 (Actual); Primary Completion 2022-09-20 (Actual); Study Completion 2022-10-20 (Actual)

PRIMARY OUTCOMES:
Change in pain. | Change in pain levels over the 10 minute session (In all three groups)
  Neonatal Pain and Stress Rating Scale; It was developed by Lundqvist et al. in 2014 to assess pain and stress in premature and newborns. The scale was adapted into Turkish by Ceylan and Bolışık (2017). It is a 3-point Likert-type scale consisting of 5 items: newborn's facial expression, breathing pattern, tone of the extremities, hand and foot activities, and activity level. Measurements are made by observation. As the score obtained increases, stress and pain increase. As a result of the evaluation, 3-5 points indicate the presence of mild pain and stress, and more than 5 points indicate the presence of severe pain and stress. The Cronbach's alpha coefficient of the scale was reported as 0.95.
Change in stress. | Change in stress levels over the 10 minute session (In all three groups)
  Neonatal Pain and Stress Rating Scale; It was developed by Lundqvist et al. in 2014 to assess pain and stress in premature and newborns. The scale was adapted into Turkish by Ceylan and Bolışık (2017). It is a 3-point Likert-type scale consisting of 5 items: newborn's facial expression, breathing pattern, tone of the extremities, hand and foot activities, and activity level. Measurements are made by observation. As the score obtained increases, stress and pain increase. As a result of the evaluation, 3-5 points indicate the presence of mild pain and stress, and more than 5 points indicate the presence of severe pain and stress. The Cronbach's alpha coefficient of the scale was reported as 0.95.
Change in behavior. | Change in behaviors over the 10 minute session (In all three groups)
  Anderson Behavioral State Scoring System-ABSS; In ABSS, which is a behavior scoring system that evaluates newborn behavior in 4 categories (eyes closed, eyes half-opened, eyes open and eyes open or closed) and 12 sub-categories, infant behaviors are scored from 1 to 12. As the score increases, it is accepted that the baby's behavior deteriorates.

CONTACTS AND LOCATIONS:
Overall Officials: Öznur BAŞDAŞ, PhD, Study Chair — TC Erciyes University
Locations (1):
- Erciyes University, Kayseri, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No